CLINICAL TRIAL: NCT00168233
Title: Impact of HIV Infection and Treatment With Highly Active Antiretroviral Therapy on Reverse Cholesterol Transport
Brief Title: Impact of HIV and Its Treatment on Reverse Cholesterol Transport
Status: Completed | Type: Observational
Sponsor: The Alfred (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Jennifer Hoy, Professor Jennifer Hoy, The Alfred
Other Study IDs: 54/05
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: HIV Infections
Keywords: Treatment Naive; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: No antiretroviral therapy for 12 months
- 2: Initiating ARV therapy with an NNRTI based regimen
- 3: Initiating ARV therapy with a PI based regimen

SUMMARY:
To investigate the effect of treatment of HIV infection with highly active antiretroviral therapy on individual steps of reverse cholesterol transport, endothelial function and intima-media thickness in HIV patients.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with HIV infection (3 groups of 50 patients each)
* HIV infected patients, naïve to ARV therapy and not likely to need to commence therapy for the duration of follow-up (12 months)
* HIV-infected patients, PI naïve, initiating therapy with PI-containing HAART (ARV naïve or NNRTI experienced changing to PI regimen)
* HIV-infected patients naïve to ARV therapy, initiating NNRTI-containing regimen

Exclusion criteria

* Treatment with any form of lipid lowering drugs, including fish oils.
* Body Mass Index greater than 27.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients naive to ARV therapy
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2005-06; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Sviridov, Dr, Study Director — Baker Heart Research Institute, Commercial Road, Melbourne; Jennifer Hoy, A/Prof, Principal Investigator — Alfred Hospital, Melbourne, Vic 3004
Locations (1):
- Alfred Hospital and Baker Heart Research Institute, Melbourne, Victoria, Australia